CLINICAL TRIAL: NCT06433089
Title: Effect of Thoracic Paravertebral Nerve Block on Postoperative Pain After Transapical Beating-heart Myectomy(TA-BSM) in Patients With Hypertrophic Obstructive Cardiomyopathy: a Retrospective Cohort Study
Brief Title: Postoperative Pain for Patients After TA-BSM
Status: Completed | Type: Observational
Sponsor: Wenlong Yao (101480) (Other)
Responsible Party: Sponsor-Investigator, Wenlong Yao (101480), Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJMZK230601
Record Dates: First submitted 2024-05-11; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Nerve Block; Transapical Beating-heart Septal Myectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group GA+PVB: The patients received General Anesthesia(GA) combined with Paravertebral Block(PVB).
  Interventions: Procedure: Thoracic paravertebral block
- group GA only: The patients received general anesthesia only.

INTERVENTIONS:
Procedure: Thoracic paravertebral block — Thoracic paravertebral block was performed before surgery
  Groups: group GA+PVB

SUMMARY:
To retrospectively analyze the intraoperative and postoperative status of patients with hypertrophic cardiomyopathy undergoing TA-BSM, and to estimate whether paravertebral nerve block can improve postoperative pain for these patients.

DETAILED DESCRIPTION:
Since conventional septal myectomy can be only assessed when the heart resumes beating, and the complications induced by cardiopulmonary bypass are inevitable, a novel transapical beating-heart septal myectomy (TA-BSM) has been invented, which provides real-time evaluation to guide resection while reducing surgical trauma. Postoperative pain after TA-BSM is unknown. Whether paravertebral nerve block can improve postoperative pain caused by TA-BSM is the objective of our study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~75 years
* American society of anesthesiologists classification II-III
* Elective TA-BSM was performed

Exclusion Criteria:

* Underwent multiple surgical procedures or required cardiopulmonary bypass assistance
* Combined other function decompensation disease
* Patients with incomplete medical records

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The information of all patients with hypertrophic cardiomyopathy undergoing TA-BSM in our hospital from April 2023 to September 2023 was extracted and screened according to the inclusion criteria and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | During the first 48 hours after surgery
  Cumulative morphine consumption

SECONDARY OUTCOMES:
Postoperative pain score 1 | 24 hours after surgery and and 48 hours after surgery
  Visual Analogue Scale score(0-10 stands for the degree of pain, 0=no pain, 10=the worst pain ever)
Postoperative pain score 2 | Day 7 after surgery and month 3 after surgery
  Brief Pain Inventory(The degree of pain [0 no pain to 10 very painful] and the impact of pain on daily life function [0 no impact to 10 very impact])
Physical recovery after surgery | Day 7 after surgery
  Quality of recovery(Rating from 0 [very poor] to 150 [excellent])
Complications | 24 hours and 48 hours after surgery
  The incidence of nausea and vomiting
Perioperative information 1 | Immediately after the surgery
  The usage of analgesic drug
Perioperative information 2 | P1= before induction, P2= 5 minutes after tracheal intubation, P3= before skin incision, P4= 5 minutes after skin incision, P5=5 minutes after placed the rib spreader
  Mean arterial blood pressure
Perioperative information 3 | P1= before induction, P2= 5 minutes after tracheal intubation, P3= before skin incision, P4= 5 minutes after skin incision, P5=5 minutes after placed the rib spreader
  Heart reat
Perioperative information 4 | Immediately after the surgery
  Duration of anesthesia
Postoperative information 1 | Postoperative in 24 hours
  Extubation time
Postoperative information 2 | Postoperative in 48 hours
  The usage of analgesic drug

CONTACTS AND LOCATIONS:
Overall Officials: Wenlong Yao, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong Science and Technology University, Wuhan, Hubei, China